CLINICAL TRIAL: NCT03834610
Title: Daily Oral L-arginine Plus Tadalafil in Diabetic Patients With Erectile Dysfunction: A Double-blinded Randomized Controlled Clinical Trial
Brief Title: Daily Oral L-arginine Plus Tadalafil in Diabetic Patients With Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Moustafa A. El Taieb, Ass. Prof. of Dermatology, Venereology and Andrology, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: L-arginine
Record Dates: First submitted 2019-02-05; First posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; Diabetes; Tadaladil; L-arginine
MeSH Terms: conditions — Erectile Dysfunction; Diabetes Mellitus | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Active Comparator): receive L-arginine 5 g oral caps daily for 8 weeks serum testosterone level measurement penile doppler
  Interventions: Drug: L-arginine 5 gm oral caps; Diagnostic Test: serum testosterone level; Diagnostic Test: HbA1C; Device: penile doppler
- Group B (Active Comparator): receive tadalafil 10 mg oral tablets daily for 8 weeks serum testosterone level measurement penile doppler
  Interventions: Drug: Tadalafil 10 MG; Diagnostic Test: serum testosterone level; Diagnostic Test: HbA1C; Device: penile doppler
- Group C (Active Comparator): receive L-arginine 5 g oral caps plus tadalafil 10 mg oral tablets daily for 8 weeks serum testosterone level measurement penile doppler
  Interventions: Drug: L-arginine 5 gm oral caps; Drug: Tadalafil 10 MG; Diagnostic Test: serum testosterone level; Diagnostic Test: HbA1C; Device: penile doppler
- Group D (Placebo Comparator): receive oral methyl cellulose daily for 8 weeks serum testosterone level measurement penile doppler
  Interventions: Diagnostic Test: serum testosterone level; Diagnostic Test: HbA1C; Device: penile doppler

INTERVENTIONS:
Drug: L-arginine 5 gm oral caps — oral L-arginine 5 gm daily for 8 weeks
  Arms: Group A; Group C
Drug: Tadalafil 10 MG — oral daily tadalafil 10mg for 8 weeks
  Arms: Group B; Group C
Diagnostic Test: serum testosterone level — measurement of serum testosterone level
Diagnostic Test: HbA1C — measurement of HbA1C levels
Device: penile doppler — penile doppler to measure the degree of erection and penile vasculature

SUMMARY:
Tadalafil is an effective oral therapy in erectile dysfunction. L-arginine is a pro drug that increase the level of nitrous oxide in the smooth muscles so can increase the strength and duration of erection. this clinical trials compare the daily oral L-arginine plus tadalafil in treatment of erectile dysfunction in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 DM

Exclusion Criteria:

* Patients with history of pelvic trauma, major pelvic surgical intervention, hypogonadism, hyperprolactinemia, hypertension, chronic prostatitis, chronic liver disease, smokers, history of chronic intake of CNS or anti-androgen drugs and patients with Peyronie's Disease or any fibrotic anomalies

Ages: 35 Years to 56 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
International Index of Erectile Function score (IIEF-5) improvement after treatment. IIEF-5 score of 22-25: No erectile dysfunction (ED), 17-21: Mild ED, 12-16: Mild to moderate ED, 8-11: Moderate ED, 5-7: Severe ED. | 8 weeks of treatment
  Efficacy of oral L-arginine 5 g plus oral tadalafil 10 mg in treatment of erectile dysfunction in diabetic patients is evaluated by International Index of Erectile Function score (IIEF-5).
Increase in Serum Total testosterone level in (nmol/L) after treatment. | 8 weeks of treatment
  Measurement of total testosterone level in (nmol/L) improvement after treatment
Improvement in Penile Doppler parameters after treatment including peak systolic velocity in (cm/sec), end diastolic volume in (cm/sec) and resistive index (RI) that = (peak systolic velocity - end diastolic velocity ) / peak systolic velocity. | 8 weeks of treatment
  Measurement of penile doppler parameters improvement after treatment peak systolic velocity in (cm/sec), end diastolic volume in (cm/sec) and resistive index (RI).

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa M El Taieb, MD, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No